CLINICAL TRIAL: NCT03766815
Title: Effect of Branched-chain Amino Acid Supplementation on Muscle Damage in Recreational Athletes
Brief Title: Effect of Branched-chain Amino Acid Supplementation on Muscle Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 113281
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Muscle Damage

STUDY DESIGN:
Intervention Model Description: Participants will be supplemented for 18 days with either 200mg BCAA/kg/day, 400mg BCAA/kg/day or placebo (fiber supplement) in jelly in a single-blind fashion. Followed by a muscle damaging exercise and subsequent MVC and blood sample for force and metabolite measurements.
Who Masked: Participant
Masking Description: Participants will not be able to distinguish branched-chain amino acid and fiber supplement by taste, color or scent as the supplements are provided in jelly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Fiber supplement mixed with jelly will be ingested for 18 days with participants performing elbow eccentric contractions as a muscle damaging exercise on the 12th-day of supplementation.
  Interventions: Dietary Supplement: Placebo; Behavioral: Muscle damaging exercise
- BCAA 200mg/kg/day (Experimental): Branched-chain amino acid supplement mixed with jelly will be ingested for 18 days. The amount of supplement provided will be based on body weight (200mg/kg/day) with participants performing elbow eccentric contractions as a muscle damaging exercise on the 12th-day of supplementation.
  Interventions: Dietary Supplement: BCAA 200mg/kg/day; Behavioral: Muscle damaging exercise
- BCAA 400mg/kg/day (Experimental): Branched-chain amino acid supplement mixed with jelly will be ingested for 18 days. The amount of supplement provided will be based on body weight (400mg/kg/day) with participants performing elbow eccentric contractions as a muscle damaging exercise on the 12th-day of supplementation.
  Interventions: Dietary Supplement: BCAA 400mg/kg/day; Behavioral: Muscle damaging exercise

INTERVENTIONS:
Dietary Supplement: BCAA 200mg/kg/day — BCAA supplement based on 200mg/kg/day for 18 days.
  Arms: BCAA 200mg/kg/day
Dietary Supplement: Placebo — Fiber supplement jelly for 18 days.
  Arms: Placebo
Dietary Supplement: BCAA 400mg/kg/day — BCAA supplement based on 400mg/kg/day for 18 days.
  Arms: BCAA 400mg/kg/day
Behavioral: Muscle damaging exercise — Participants will be asked to perform muscle damaging elbow eccentric contraction exercise at 120% of 1RM for three sets of 15 repetitions with the dominant arm at maximal effort on a Biodex machine with a 3 minute rest period between each set.

SUMMARY:
Seventy-eight recreational athletes who never resistance trained will be randomly assigned into three groups of twenty-six. Branched-chain amino acid will be supplemented for 18days at 0, 200 or 400 mg/body weight(kg)/day in jelly. Participants will be asked to perform elbow flexions on the 12th day of supplementation. Maximum voluntary contractions will be measured before, during and after the supplementation period to compare the effects of different doses of branched-chain amino acid has on muscle damage markers.

DETAILED DESCRIPTION:
Previous studies have not been able to show consistent effects due to various reasons. The major limitations are the lack of enough data on the amount and duration of branched-chain amino acid supplementation, and the level of muscle damage for branched-chain amino acid to be effective. Based on a recent meta-analysis, it has been suggested that to be effective, branched-chain amino acid should be supplemented more than 200mg/kg/day before a low-to-moderate intensity exercise bout. Therefore, this study is designed based on the above suggestions and to compare the effect of different doses of branched-chain amino acid on muscle damage markers in healthy recreational active individuals.

Three treatment groups (n=26) will be randomly assigned to be supplemented with either 200mg BCAA/kg/day (BCAA200), 400mg BCAA/kg/day (BCAA400) or placebo (fiber supplement; PL). Supplements will be provided in jelly in a single blind fashion to be ingested 1hour after each of the three main daily meals for 18days. Anthropometric measurements (body weight, lean mass, height), body temperature, ultrasound (US), strength assessment (maximal voluntary contraction, MVC), resting metabolic rate (RMR), rate of perceived exertion (RPE), delayed onset of muscle soreness (DOMS) and blood samples (duplicates; myoglobin; BCAA) will be collected before, during and after the supplementation period at different time points (see appendix for the above tables). Repeated-bout effect (RBE) on both arms will be measured 7 days after the damage inducing session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females at the age of 18-40
* Endurance trained athletes
* Weekly exercise duration is less than 150minutes but more than 30 minutes

Exclusion Criteria:

* Individuals who cannot endure three days for not eating meat
* Diabetic
* Have been performing resistance trainings
* Have been taking protein supplement
* Have been consuming a high level of protein in the regular diet
* Have been taking omega-three and vitamin E supplements
* Have been taking anabolic Steroids
* Have been taking regular medications
* Have cardiovascular Disease
* Have a history of joint & Muscle Injuries
* Females with irregular Menstrual Cycle

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximum voluntary contraction (MVC) | baseline (before supplementation) and at 1,3,24,48,72,96,120,144 hours after muscle damage
  Participants will be asked to perform three repetitions of concentric elbow flexion at their maximal force (1RM) with both their dominant and non-dominant arm on an isokinetic dynamometer (Biodex).

SECONDARY OUTCOMES:
Change in blood myoglobin | 10 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Blood myoglobin will be measured with Enzyme-Linked Immunosorbent Assay.
Change in 3-methyl-histidine | 10 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Ultra-performance liquidchromatography tandem mass spectrometry (UPLC-MS/MS) using an Acquity Ultra Performance LC system coupled to a Waters Quattro Premier XE mass spectrometer (bothWaters Corporation, Milford, MA, USA) and the Waters MassLynx Software (Version 4.1).
Changes in insulin | 10 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Blood insulin will be measured with a standard insulin radioimmunoassay kit.
Change in muscle soreness | 10 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Perceived muscle soreness will be determined by asking participants to stand in the anatomical position while flexing the shoulder of the exercised arm at 90degrees and fully extending the elbow. Participants will be asked to determine their forearm flexor muscles soreness with the use of a visual analogue scale (VAS) and rate from 1 being no pain and 10 being extremely painful.
Change in ultrasound images of the arm muscles | 10 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Ultrasound measurements will be used to scan the triceps brachii and the forearm flexors. A permanent marker will be used to mark the elbow joint as the origin and both the belly of the triceps and the belly of the flexor digitorum profundus as the end point so as to compare the echoic difference in both the upper and lower arms.
Change in limb girth | 10 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Limb girth of the upper arm (between the lateral epicondyle of the humerus and the acromion process) and the lower arm (between the lateral epicondyle of the humerus and the styloid process of the radius) will be measured with an anthropometric tape when the arm is naturally hanging down.
Change in body temperature | 20 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Body temperature will be measured with an ear thermometer
Change in resting metabolic rate | 20 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Resting metabolic rate will be measured with a metabolic cart
Change in range of motion | 20 min before muscle damaging exercise and at each of 1,3,24,48,72,96,120,144 hours after muscle damage
  Range of motion of the arm will be measured by asking the participant to stand in the anatomical position while fully flexing the shoulder of the exercised arm and then extending the elbow to an angle that they do not feel any pain in the arms. A goniometer will be used to measure the angles.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No